CLINICAL TRIAL: NCT02584517
Title: Understanding the Aetiology and Pathogenesis of Giant Cell Arteritis
Brief Title: Aetiology of TemporaL Arteritis Study
Acronym: ATLAS
Status: Withdrawn | Type: Observational
Why Stopped: Lack of funding
Sponsor: University of Oxford (Other)
Collaborators: University of Leeds (Other)
Responsible Party: Sponsor
Other Study IDs: ATLAS001
Record Dates: First submitted 2015-10-21; First posted 2015-10-22 (Estimated); Last update posted 2022-08-15 (Actual); Status verified 2015-10

CONDITIONS: Temporal Arteritis
Keywords: Vasculitis; Autoimmune disease; Connective tissue disease; Polymyalgia rheumatica; Musculoskeletal Diseases; Immune disorder; Rheumatic disease
MeSH Terms: conditions — Giant Cell Arteritis; Vasculitis; Autoimmune Diseases; Connective Tissue Diseases; Polymyalgia Rheumatica; Musculoskeletal Diseases; Immune System Diseases; Rheumatic Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum Plasma Peripheral Blood Mononuclear Cells Whole blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- GCA: Patients referred with suspected GCA, whose final diagnosis is GCA
- Not GCA: Patients referred with suspected GCA, whose final diagnosis is another disorder

SUMMARY:
Giant Cell Arteritis (GCA) is the most common vasculitis and has significant morbidity in terms of blindness, stroke, and tissue necrosis. It requires protracted treatment with high-dose steroids, and despite this there is a risk of flare during the treatment. Little is known about the initial triggers for the inflammatory process, and there are no good markers of response or relapse. We will study patients referred with suspected GCA to identify important components of the immune response in GCA, and follow them over time to collect evidence of how best to monitor their condition.

DETAILED DESCRIPTION:
Objectives and Study Plan:

Study Purpose:

The purpose of the study is to investigate the underlying immunological processes in GCA and to study the pattern of expression of immune response over time to give us information about how best to monitor GCA.

End Point:

The end point will be the final visit of the final patient.

Milestones:

The project is in 3 phases. In phase 1 (0-2 years) patients will be recruited to fulfil the specified primary and secondary objectives. In phase 2 (0-4 years), these patients will be followed up for a total of 2 years each, or until they are discharged from clinic. In phase 3 (1-5 years), further studies will be defined and tissue and data collected under amended ethics.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or over
2. A clinical suspicion of a new diagnosis of GCA e.g. patients with a new onset of headache, scalp tenderness, with or without elevated CRP or ESR, jaw or tongue claudication with or without visual loss
3. Participants must be willing to give informed written consent or willing to give permission for a nominated friend or relative to provide written informed assent if they are unable to do so because of physical disabilities e.g. sudden onset of blindness/vision loss which can be caused by GCA (this will be made clear in the ethics approval application)

Exclusion Criteria:

1. Previous diagnosis of GCA
2. Long term (>1 month) high dose (>20mg per day at any time) steroids for conditions other than PMR, within three months prior to study entry
3. Inability to give informed consent (either written consent or verbal assent from a relative or carer)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The proposed study will recruit a cohort of eligible patients (predominantly from primary care referrals) suspected by their referring doctor to have new onset of GCA.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2016-01; Primary Completion 2018-01 (Estimated); Study Completion 2021-01 (Estimated)

PRIMARY OUTCOMES:
Phenotyping of innate lymphoid cells (ILC) in the arterial wall and blood of patients with GCA | 24 months
  Arterial biopsy tissue and peripheral blood will be collected from patients with suspected GCA. A proportion of these will be diagnosed with GCA and will be the "test" subjects, and a proportion will be diagnosed with other conditions that are not GCA and will be the "controls". We will use immunohistochemistry and immunofluorescence microscopy to locate and phenotype ILC in arterial biopsies. We will use semi-quantitative methods (ie cells per random high powered field) to compare prevalence of ILC in tests and controls. We will also isolate peripheral blood mononuclear cells (PBMCs) from fresh whole blood, and stain the cells to use flow cytometry to quantify and phenotype the ILC. Tests and Controls will be compared using Mann-Whitney statistical testing.

SECONDARY OUTCOMES:
CD70 in GCA | 12 months
  CD70 is a costimulatory molecule which is present for a short time on the surface of activated T cells. CD70 has been studied in other autoimmune conditions such as systemic lupus, where it is involved in generating the self-reactive factors responsible for the disease. It is therefore suggested that it might be involved in the development of another autoimmune vasculitis, GCA. We will quantify and phenotype CD70+ve cells in peripheral blood and biopsies of patients with GCA and in controls. We will also measure the levels of the soluble form of its receptor, CD27, in patients and controls.
IL-7 and sIL-7R in GCA | 36 months
  IL-7 is a key cytokine for development of all lymphoid cells, including ILC. Levels of sIL-7R have been linked to active renal disease in systemic lupus, and sIL-7R is suggested as a biomarker of lupus. We will collect serum at several time points from patients with GCA and controls (see primary outcome measures). The level of IL-7 and sIL-7R will be quanitified by Enzyme-linked Immunosorbent Assay (ELISA) and the results plotted as time series. We will analyse the trends of these series to see how useful IL-7 and sIL-7R may be in monitoring GCA.
Vascular Endothelial Growth Factor (VEGF) levels over time | 36 months
  VEGF is a putative biomarker of GCA. We will collect serum at several time points from patients with GCA and controls (see primary outcome measures). The level of VEGF will be quanitified by Enzyme-linked Immunosorbent Assay (ELISA) and the results plotted as time series. We will analyse the trends of these series to see how useful VEGF may be in monitoring GCA.
Pentraxin 3 levels over time | 36 months
  Pentraxin 3 is a second biomarker of interest in GCA, and we plan to analyse its expression in peripheral blood as for VEGF.
Archiving of tissue for future studies | 60 months+
  The cohort of patients recruited to this study represents a valuable resource for future ethically-approved studies of the aetiology of GCA. We believe that the majority of patients would like their donations to contribute to as much research as possible. Therefore we will archive tissue in the form of blood fractions and temporal artery biopsy specimens, as well as linking to anonymized clinical and imaging data. It is planned that the study ethics will be amended with novel substudies as they are designed.

CONTACTS AND LOCATIONS:
Overall Officials: Raashid A Luqmani, DM FRCP, Principal Investigator — University of Oxford

REFERENCES:
- [Result] Weyand CM, Goronzy JJ. Immune mechanisms in medium and large-vessel vasculitis. Nat Rev Rheumatol. 2013 Dec;9(12):731-40. doi: 10.1038/nrrheum.2013.161. Epub 2013 Nov 5. PMID 24189842
- [Result] Artis D, Spits H. The biology of innate lymphoid cells. Nature. 2015 Jan 15;517(7534):293-301. doi: 10.1038/nature14189. PMID 25592534
- [Result] Ciccia F, Guggino G, Rizzo A, Saieva L, Peralta S, Giardina A, Cannizzaro A, Sireci G, De Leo G, Alessandro R, Triolo G. Type 3 innate lymphoid cells producing IL-17 and IL-22 are expanded in the gut, in the peripheral blood, synovial fluid and bone marrow of patients with ankylosing spondylitis. Ann Rheum Dis. 2015 Sep;74(9):1739-47. doi: 10.1136/annrheumdis-2014-206323. Epub 2015 Apr 22. PMID 25902790
- [Result] Kozlowska A, Hrycaj P, Lacki JK, Jagodzinski PP. Fyn and CD70 expression in CD4+ T cells from patients with systemic lupus erythematosus. J Rheumatol. 2010 Jan;37(1):53-9. doi: 10.3899/jrheum.090424. Epub 2009 Dec 1. PMID 19955046
- [Result] Lauwerys BR, Husson SN, Maudoux AL, Badot V, Houssiau FA. sIL7R concentrations in the serum reflect disease activity in the lupus kidney. Lupus Sci Med. 2014 Jul 17;1(1):e000036. doi: 10.1136/lupus-2014-000036. eCollection 2014. PMID 25396066